CLINICAL TRIAL: NCT02890732
Title: Implementation and Evaluation of a Prototype Smartphone Application of Personalized Care of Patients After Hospitalization for Coronary Artery Disease
Brief Title: Evaluation of a Prototype Smartphone Application of Personalized Care for Coronary Artery Disease
Acronym: AppET-Coeur
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7417
Record Dates: First submitted 2016-07-20; First posted 2016-09-07 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Appet HEART (Experimental): smartphone application prototype of personalized care of patients after hospitalization for coronary artery disease
  Interventions: Device: Appet HEART

INTERVENTIONS:
Device: Appet HEART — smartphone application prototype of personalized care of patients after hospitalization for coronary artery disease

SUMMARY:
This project will benefit from the results of the concept study conducted from July to October 2014 from groups of coronary patients. This first study will help to develop the precise contours of Appet HEART application for the production of the prototype version used in the clinical feasibility study.

The objectives of the feasibility study are:

1. assess the rate of use of the application
2. to determine the ideal target population of the application
3. to evaluate the effectiveness of the application
4. to measure the risks and potential limitations of its use
5. to determine the medical and economic impact of this application

DETAILED DESCRIPTION:
The patient education activities at the center in coronary artery disease, and have shown their efficiency, in combination with exercise training. Unfortunately the issue of educational care is low and maintaining long-term changes in the lifestyle and adherence to drug intake is limited which is a major health challenge because originally a recidivism rate too high coronary disease. In this context, therapeutic measures to enable patients to better integrate into their daily lives the recommendations in the long term are fundamental.

As part of the expertise of the Toulouse University Hospital in the field of therapeutic education coronary patient, the investigators decided to develop a Smartphone application that aims to strengthen and modernize the educational care to the patient. Based on an accurate and comprehensive assessment of lifestyle, from the technical elements of Smartphone support, but also on providing innovative educational materials (videos, interactive software...), the treat ( pharmacological or not: diet, physical activity, toxic consumption ) may thus be optimized according to the principle of telemedicine.

This project will benefit from the results of the concept study conducted from July to October 2014 from groups of coronary patients. This first study will help to develop the precise contours of Appet HEART application for the production of the prototype version used in the clinical feasibility study.

The objectives of the feasibility study are:

1. assess the rate of use of the application
2. to determine the ideal target population of the application
3. to evaluate the effectiveness of the application
4. to measure the risks and potential limitations of its use
5. to determine the medical and economic impact of this application

This is a single-center study. Patients will be recruited from the Toulouse University Hospital in cardiac services when patients came to coronary heart disease. After inclusion, patients receive an initial educational diagnosis that will determine individualized educational goals on the management of their coronary disease. Patients then receive training in the use of Appet HEART application. Using the application is provided on year.

The evaluation criteria of the study is original because conducted in hetero or self during the protocol monitoring time. Chronologically the investigators note:

* An initial assessment hetero judgments criteria
* A self- evaluation every three months for one year via their smartphone on some of these criteria via questionnaires
* A final visit is scheduled to perform the same hetero- evaluation at the initial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary heart disease aged 18 to 80 years, from an therapeutic patient education in Cardiology, capable of using a Smartphone application and with a Smartphone

Exclusion Criteria:

* Disorders of understanding, lack of long-term conditions, legal protection measure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hours ou use per patient per month | 12 months
  Hours of use of the new smartphone application per patient per month

CONTACTS AND LOCATIONS:
Overall Officials: Marc Labrunee, Dr, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Yes